CLINICAL TRIAL: NCT00081991
Title: A Cross Sectional Clinical Study of Human Lens Aging and Cataract Formation, in Vivo, Using Dynamic Light Scattering (DLS)
Brief Title: Dynamic Light Scattering for Studying Lens Aging and Cataract Formation
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040166; 04-EI-0166
Record Dates: First submitted 2004-04-28; First posted 2004-04-28 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-04

CONDITIONS: Cataract
Keywords: Cataract; Blindness; Clinical; Human Aging; Dynamic Light Scattering (DLS); Aging-Related Lens Changes; Early Cataract; Lens; AREDS Grading; In Vivo; Healthy Volunteer
MeSH Terms: conditions — Cataract; Blindness

SUMMARY:
This study will use dynamic light scattering (DLS) technology to study normal lens aging and early cataract formation. Cataract is a clouding of the lens that interferes with the passage of light to the retina, impairing visual acuity. DLS uses a low intensity laser light (similar to that used in supermarket checkouts) to measure lens cloudiness. It detects changes in the human lens at the earliest molecular stages of cataract development, when anti-cataract treatment would be most effective in reversing, delaying or preventing cataract formation.

Healthy normal volunteers and patients with age-related cataract between 18 and 80 years of age may be eligible for this study. Participants undergo the following tests and procedures:

Medical history

Eye examination, including the following:

* Measurement of visual acuity (vision chart)
* Measurement of eye pressure
* Dilation of the pupils for slit lamp (microscope) examination and grading of lens opacity
* Ultrasound examination of the eye to determine distances between cornea, lens (including lens thickness), and retina
* Examination of the retina at the back of the eye
* Dynamic light scattering of the lens (see below)
* Lens photography using a camera with a bright flash

For the DLS procedure, the patient sits in front of the DLS device with his or her chin placed on a chin rest and fixes on a yellow target in the center of the camera lens. When the eye is properly aligned, DLS measurements are taken on the lens.

DETAILED DESCRIPTION:
A new non invasive, in vivo technique to study the molecular changes in the human lens, called Dynamic Light Scattering Device (DLS), has recently been developed. Preliminary studies have shown its potential to detect the earliest changes in cataract, at the stage where anti-cataract treatment would be most effective in reversing, delaying or preventing cataracts. A new miniaturized version of this device has been developed by NASA using lower energy lasers, and under a NASA-NEI Inter Agency Agreement, has been successfully developed into a clinical device at the NEI. We recently conducted pilot studies to evaluate the usefulness and reproducibility of this instrument for quantitating human lens changes, and found good reproducibility. We also derived a useful parameter to use with this new technique, the log mean particle size, derived from particle size distribution data. Preliminary studies have also shown that the NASA-NEI DLS device can be used to detect and monitor molecular changes in early cataract formation as well as in normal aging. We therefore propose to conduct a larger cross sectional clinical study to detect and monitor molecular changes in the lens in early cataract formation and in normal aging.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients aged 18-80 years will be admitted to this study. There will be no racial or gender bias in the recruitment.

227 patients with AREDS nuclear cataract grades 2 or less will be enrolled in the study. 40 patients with AREDS nuclear cataract grade 3 and 4 will also be enrolled.

For those patients enrolled in the study, both eyes will be evaluated for this protocol. However, the participant has the right to choose to undergo measurements only in one eye. In that case, the eye to be examined will be determined by the partipantt's birth month. If the patient's birth month is an even number, the right eye will be examined; if the patient's birth month is odd, the left eye will be examined.

EXCLUSION CRITERIA:

Subjects who have tear film disorders, corneal opacities or disorders, uveitis, glaucoma or who have difficulty fixating, will be excluded.

Subjects who are thought to be at risk for an adverse reaction to pupil dilation, or have a history of allergic reaction to one of the dilating agents that will be used, will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 267
Dates: Start 2004-04; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Benedek GB, Chylack LT Jr, Libondi T, Magnante P, Pennett M. Quantitative detection of the molecular changes associated with early cataractogenesis in the living human lens using quasielastic light scattering. Curr Eye Res. 1987 Dec;6(12):1421-32. doi: 10.3109/02713688709044506. PMID 3427992
- [Background] Datiles M, Podgor M, Edwards P. Reproducibility of the Early Cataract Detector (Kowa ECD 2000). Ophthalmic Surg. 1988 Sep;19(9):664-6. PMID 3186178
- [Background] Bursell SE, Baker RS, Weiss JN, Haughton JF, Rand LI. Clinical photon correlation spectroscopy evaluation of human diabetic lenses. Exp Eye Res. 1989 Aug;49(2):241-58. doi: 10.1016/0014-4835(89)90094-8. PMID 2767171